CLINICAL TRIAL: NCT01126762
Title: A Pilot Randomized Controlled Trial to Promote Healthful Fish Consumption in Pregnancy
Brief Title: Trial of Fish Intake Advice in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Harvard University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Emily Oken, Associate Professor, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPHCI Fish 0344; P30ES000002 (NIH); P30DK040561 (NIH); R01ES016314 (NIH); K24HD069408 (NIH)
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Nutrition
Keywords: Docosahexaenoic acid; fish; pregnancy; methylmercury; n-3 polyunsaturated fatty acid
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dietary advice and grocery store card (Experimental): Dietary advice to consume low mercury, high DHA fish plus a grocery store gift card to support the purchase of fish
  Interventions: Behavioral: Dietary advice
- Dietary advice (Experimental): Dietary advice regarding consumption of low mercury, high DHA fish
  Interventions: Behavioral: Dietary advice
- Control (Placebo Comparator): General dietary advice not focused on fish intake
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Dietary advice — Dietary advice regarding consumption of low mercury, high DHA fish
  Arms: Dietary advice; Dietary advice and grocery store card
Behavioral: Control — Advice regarding healthful diet during pregnancy, not focused on fish intake
  Arms: Control

SUMMARY:
The overall goal of this project is to establish a pilot study to develop and refine an intervention to promote consumption of fish low in mercury and high in n-3 PUFA among pregnant women. The investigators will demonstrate our ability to recruit pregnant women, influence their fish consumption, and measure changes in nutrient and toxicant biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* Currently pregnant 12-22 weeks
* Singleton pregnancy
* Consuming fish <=2 times per month

Exclusion Criteria:

* Inability to answer questionnaires in English
* Plans to leave study area prior to delivery
* Would never eat fish (e.g. vegan, allergy to fish)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Plasma elongated n-3 PUFA levels | 12 weeks
  Change in plasma levels of elongated n-3 PUFA from recruitment to follow up at 12 weeks

SECONDARY OUTCOMES:
Whole blood mercury | 12 weeks
  Change in whole blood total mercury level from recruitment to 12 weeks
Fish consumption | 12 weeks
  Change in fish consumption from recruitment to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emily Oken, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (1):
- Harvard Pilgrim Health Care, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Oken E, Guthrie LB, Bloomingdale A, Gillman MW, Olsen SF, Amarasiriwardena CJ, Platek DN, Bellinger DC, Wright RO. Assessment of dietary fish consumption in pregnancy: comparing one-, four- and thirty-six-item questionnaires. Public Health Nutr. 2014 Sep;17(9):1949-59. doi: 10.1017/S1368980013001985. Epub 2013 Jul 24. PMID 23883550
- [Derived] Oken E, Guthrie LB, Bloomingdale A, Platek DN, Price S, Haines J, Gillman MW, Olsen SF, Bellinger DC, Wright RO. A pilot randomized controlled trial to promote healthful fish consumption during pregnancy: the Food for Thought Study. Nutr J. 2013 Mar 15;12:33. doi: 10.1186/1475-2891-12-33. PMID 23496848